CLINICAL TRIAL: NCT02299115
Title: Prednisolone vs. Vigabatrin in the First-line Treatment of Infantile Spasms
Brief Title: Prednisolone Versus Vigabatrin in the First-line Treatment of Infantile Spasms
Acronym: PREDVGB
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Most centres are now using oral steroids as 1st line treatment so question of efficacy is no longer of high interest.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Carter Snead, Staff Neurologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000045463
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Infantile Spasms
Keywords: Vigabatrin; Prednisolone
MeSH Terms: conditions — Spasms, Infantile | interventions — Prednisolone; Vigabatrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone (Experimental): Single center, prospective, observational, open trial using high-dose oral prednisolone as first-line treatment for newly diagnosed Infantile Spasms (non-Tuberous Sclerosis)
  Interventions: Drug: Prednisolone
- Vigabatrin (Active Comparator): Retrospective controls composed of our cohort of non-Tuberous Sclerosis Infantile Spasms patients from January 2010- September 2013 who received Vigabatrin as first-line treatment.
  Interventions: Drug: Vigabatrin

INTERVENTIONS:
Drug: Prednisolone — Corticosteroid
  Other Names: pms-prednisolone
  Arms: Prednisolone
Drug: Vigabatrin — Antiepileptic
  Other Names: Sabril
  Arms: Vigabatrin

SUMMARY:
Infantile Spasms, is an rare age-specific epilepsy of early infancy. A 2012 American Academy Neurology/ Child Neurology Society practice parameter update on the medical treatment of infantile spasms concluded: adrenocorticotrophic hormone or vigabatrin may be offered for short-term treatment of infantile spasms. There was insufficient evidence to recommend the use of prednisolone, dexamethasone, and methylprednisolone. The cost of ACTH and the side effects of vigabatrin have led to the consideration of alternative medications to treat infantile spasms. The United Kingdom Infantile Spasms Study (UKISS) in 2004, comparing the efficacy of intramuscular synthetic ACTH to high dose oral prednisolone, showed a response rate of 74% for ACTH and 70% for prednisolone. Since the UKISS paper was published, many institutions in the United States and Australia have used oral prednisolone instead of ACTH, partly due to the exorbitant cost of intramuscular ACTH but also its ease of use and better adverse event profile compared to ACTH. Prednisolone and vigabatrin are both oral medications, which can be initiated promptly upon diagnosis of infantile spasms, expediting treatment and shortening treatment lag time. Because the UKISS trial is the only Class 3 study providing evidence for oral prednisolone in the first-line treatment of infantile spasms, further prospective studies are needed.

DETAILED DESCRIPTION:
Background and Rationale for the study:

Infantile spasms (IS) is a rare, catastrophic age-specific epilepsy syndrome with onset within the first 12 months of life. The disorder is characterized clinically by epileptic spasms, often accompanied by developmental regression and a characteristic interictal electroencephalography (EEG) pattern called hypsarrhythmia. When all these three features are present, the term, "West syndrome" is commonly used. The catastrophic nature of the disorder is due to the frequent sequelae of severe global neurodevelopmental delay and medically refractory epilepsy.

The initial age of onset in 90% of cases occur before 12 months of life, with peak onset at 6 months. The incidence is 2 to 3 per 10,000 live births with a lifetime prevalence of 1.5 to 2 per 10,000 children. It is slightly more common in males, and a family history exists in 3%-6% of cases.1,2,3 The etiology of IS has conventionally been divided into symptomatic or cryptogenic, depending on whether the underlying cause is known. Conditions causing symptomatic IS are diverse and can include focal or multifocal brain injuries, chromosomal abnormalities and genetic mutations and inborn errors of metabolism. In about 20% of cases, the identifiable cause remains unknown and these are defined as cryptogenic.

The spontaneous remission rate of IS in limited natural history studies is 30%.4,5 Although the clinical spasms and typical EEG pattern disappear by 3 to 4 years of age, up to 60% of children with IS will go on to develop other types of refractory seizures, including Lennox Gastaut syndrome. The poor developmental outcome in IS is primarily due to the underlying etiology, however, delay in diagnosis and treatment6 and the use of ineffective therapies are also contributory factors. The hypsarrhythmia EEG pattern is a pattern of epileptic encephalopathy and there is evidence that longer duration of epileptic encephalopathy contributes to developmental delay and to the development of autism, especially in infants with Down syndrome and tuberous sclerosis complex (TSC).7,8 Currently, there is still considerable variation in the management of IS, as evidenced by the US Consensus Report and a recent survey done on the current evaluation and treatment of IS among members of the Child Neurology Society (CNS). Most neurologists use adrenocorticotrophic hormone (ACTH) as their preferred, first-line treatment of IS, not caused by TSC and Vigabatrin (VGB) as the first-line treatment of IS caused by TSC. 9,10 The 2004 American Academy of Neurology (AAN) and CNS practice parameter on the medical treatment of IS and the 2012 update of this evidenced-based guideline concluded that ACTH or VGB may be useful for the short-term treatment of IS, with ACTH being more effective than VGB excluding cases with TSC. 11,12 The 2012 update also concluded that there is insufficient evidence to determine whether other forms of corticosteroids are as effective as ACTH. There is also insufficient evidence to recommend other agents, or combination therapy in the short-term treatment of IS.

Although many conditions can cause IS, several hypotheses regarding the underlying mechanisms have been proposed. The corticotrophin releasing hormone (CRH) hypothesis is one of the most studied. Children with IS, have the common characteristic of excessive release of CRH. Elevated CRH can cause seizures and neuronal death within the hippocampus and amygdala of immature brains in animal studies. Elevated CRH also cause desensitization of CRH receptors leading to decreased ACTH release and resulting in reduced ACTH levels in the cerebrospinal fluid (CSF). ACTH treatment, most likely suppresses the excessive production of CRH via direct action on melanocortin receptors eliciting an antiepileptic effect.13 Prednisolone is a primary metabolite of a synthetic glucocorticoid, prednisone. Corticosteroids can reduce hippocampal excitability in vitro, increases gamma-aminobutyric acid (GABA) and antagonize 5-hydroxytryptophan.14 VGB is an irreversible, enzyme-activated, selective inhibitor of GABA-transaminase. By inhibiting its catabolism, there is increased availability of GABA within the synaptic cleft, increasing its inhibitory effect.15 The mammalian target of rapamycin (mTOR) pathway is a key signaling pathway that is dysregulated in TSC. Animal studies have shown that VGB partially inhibited mTOR pathway activity and glial proliferation in the knock-out mice in vitro, as well as reduced mTOR pathway activation in cultured astrocytes from both knock-out and control mice. This may account for the unique efficacy of VGB in TSC.16

At our institution, VGB is the preferred first-line treatment for all newly diagnosed IS due to its relative ease of use and fewer acute adverse events compared to ACTH. However, concerns regarding retinal toxicity17 require regular monitoring with electroretinograms (ERGs) performed under sedation.18 Also, VGB-related MRI changes are seen in 22-32% of children treated for IS and although these changes are mostly asymptomatic and may resolve even when VGB is continued, there is concern that the changes reflect a medication-related neurotoxic effect.19,20 For patients who fail VGB, we use a 6-week course of synthetic ACTH (Synacthen) given intramuscularly (IM) every other day as second-line agent. However, it is associated with significant adverse events, which include infections from immunosuppression, arterial hypertension, weight gain, severe irritability, gastric irritation, hyperglycemia, electrolyte disturbances, cerebral atrophy, and behavioral changes.

The United Kingdom Infantile Spasms Study (UKISS) demonstrated the superiority of hormonal therapy over VGB for cessation of spasms at 14 days in infants without TSC. The hormonal therapy arm included patients allocated high-dose oral prednisolone and intramuscular ACTH and the study showed that prednisolone was as effective as ACTH.21 Because this is the only Class 3 study providing evidence for oral prednisolone in the first-line treatment of IS, further prospective studies are needed.

Since 2010, the Hospital for Sick Children (SickKids) started providing the option of either IM ACTH or high-dose oral prednisolone as second-line treatments when patient failed VGB. Our previous retrospective case review of twenty IS patients who had failed a 2-week course of VGB showed an 80% response rate (12/15) to ACTH and only 20% (1/5) to prednisolone. 22. This seemingly low response to prednisolone may be due to the underlying etiology, which made the condition refractory to VGB in the first place.

Since the UKISS paper was published, many institutions in the US and Australia have used oral prednisolone instead of ACTH, partly due to the exorbitant cost of intramuscular ACTH (US$70,000 per course for natural ACTH) but also its ease of use and better adverse event profile compared to ACTH.23,24 A retrospective case series of 17 newly diagnosed IS given high-dose oral prednisolone as first-line treatment showed clinical response of 100% in the cryptogenic group, and 64% in the symptomatic (non-TSC) group.24 A retrospective case series of 27 newly diagnosed IS given high dose prednisolone (8mg/kg/day) with a maximum daily dose of 60 mg showed a 63% response rate (17/27) to prednisolone within 2 weeks. 25

The selection of the starting dose and 4 week, duration of treatment was based on the previous studies, which used a dose range of 4-8 mg/kg/day and 8mg/kg/day respectively with 4 - 6 weeks duration of therapy. 21.23.24.25.

We elected to use the higher end of the dose range previously reported to ensure maximum efficacy, with the shorter length of 4 weeks of treatment to reduce the risk of medication side effects.

The relapse rate for infantile spasms in retrospective studies has ranged between 12-40%, with time to relapse between 2-25 months. 24,25. We do not envisage using long-term treatment or recurrent intermittent treatment with prednisolone.

Prednisolone and VGB are both oral medications, which can be initiated promptly upon diagnosis of IS, expediting treatment and shortening treatment lag time. We propose that oral prednisolone may be more effective than VGB when used as a first-line treatment in newly diagnosed non-TSC IS patients.

and Objective of the study: Aim To compare the efficacy of prednisolone and VGB as 1st line short-term treatment of IS as measured by clinical and EEG response at 2 weeks.

Hypothesis:

More patients allocated to prednisolone therapy will have cessation of spasms and resolution of hypsarrhythmia at 2 weeks.

METHODS:

Study design:

Single center, prospective, observational, open trial using high-dose oral prednisolone as first-line treatment for newly diagnosed IS (non-Tuberous Sclerosis), with follow up at 2 weeks, the end of treatment and then 5 months later. All patients will undergo thorough history, physical and neurological examination, metabolic, genetic, EEG and neuroimaging studies as per the Hospital for Sick Children (HSC) Infantile Spasms Guidelines. 25 These patients will be compared to our historical controls, composed of our cohort of non-TSC IS patients from January 2010- September 2013 who received VGB as first-line treatment, met the inclusion criteria and were followed up for at least 6 months from diagnosis and treatment initiation.

The patients and their families are under no obligation to be involved in the study and will continue to receive care from their primary neurologists should they choose not to participate in the study.

Study Duration: The length of the study for each patient will be approximately 6 months. The total duration of the study is estimated at 3 years.

Sample size: A sample population of 70 patients in the retrospective VGB cohort and 35 patients in the prospective Prednisolone cohort with a 2:1 match are required to demonstrate a statistically significant difference in efficacy of 25% between Prednisolone and Vigabatrin.

Patient Population: Children between the ages of 2-24 months with a clinical spasms and hypsarrhythmia or modified hypsarrhythmia on initial EEG referred to the outpatient Neurology clinic at Sickkids.

Control Population: Historical controls will be composed of our cohort of non-TSC IS patients from 2010-2013 who received VGB as first-line treatment and fulfill the inclusion criteria for the study.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria:

1. Age 2-24 months
2. Clinical spasms
3. Initial EEG with hypsarrhythmia or modified hypsarrhythmia

The inclusion criteria do not quantify the initial severity or frequency of infantile spasms. Infantile spasms is a unique epileptic disorder characterized by clusters of brief infantile spasms, where each one lasts a few seconds and cluster may last minutes. The diagnosis of infantile spasms and response to medication depends on the presence or absence of these events and the frequency of infantile spasms has not been used to determine medication efficacy in previous studies. A seizure diary will be used to quantify the seizure burden, however efficacy will depend on complete resolution of clinical spasms and resolution of hypsarrhythmia on EEG -

Exclusion Criteria:

1. Age <2months or older than 24 months
2. Tuberous sclerosis (if known at the time of enrolment)
3. Previous treatment (within 28 days) with VGB or hormonal treatments
4. Contraindications to hormonal therapy: This includes untreated systemic fungal infections, known hypersensitivity to prednisolone or other corticosteroids, or to any of the non-medicinal ingredients present in the solution. Active or latent tuberculosis, ocular herpes simplex, hypothyroidism, hepatic cirrhosis, nonspecific ulcerative colitis, abscess or other pyogenic infection, fresh intestinal anastomoses, active or latent peptic ulcer, renal insufficiency, hypertension, osteoporosis, cardiac disease, thromboembolic disorders and diabetes mellitus. All patients with cardiac risk factors will receive an electrocardiogram (ECG), chest xray (CXR) and cardiology referral if indicated. Patients diagnosed with cardiac disorders will be excluded from the study since high dose steroids may exacerbate arrhythmias.
5. Inability of parents or guardians to give consent
6. Enrolment in a concurrent treatment trial that might affect outcome measures of this trial -

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Resolution of Infantile spasms and Hypsarrhythmia | 14 days
  Clinical response: cessation of spasms: no reported spasms for at least 48 hours including day 14 of the trial.
  EEG response: complete resolution of hypsarrhythmia or modified hypsarrhythmia pattern, on follow up EEG at approximately 2 weeks of the trial.

SECONDARY OUTCOMES:
Clinical or EEG relapse of Infantile Spasms | 6 months
  Clinical relapse: any spasm occurring after 2 weeks up to and including final clinical assessment at approximately 5 months (+/- 2weeks) post-treatment in an infant who had cessation of spasms.
  EEG Relapse: recurrence of hypsarrhythmia/modified hypsarrhythmia pattern after one previous EEG showing resolution of hypsarrhythmia
Seizure outcome at final follow up (presence or absence of any seizure types at final follow up as assessed by seizure diary and on history at final follow up visit) | 6 months
  Clinical assessment of the presence or absence of any seizure types at final follow up as assessed by seizure diary and on history at final follow up visit.
Time to cessation of Infantile spasms | 14 days
  Length of time in days to achieve cessation of Infantile spasms
Time to relapse | 6 months
  Length of time (in days) from the initial resolution of Infantile spasms to the relapse of Infantile spasms

CONTACTS AND LOCATIONS:
Overall Officials: Carter Snead, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riikonen R. Epidemiological data of West syndrome in Finland. Brain Dev. 2001 Nov;23(7):539-41. doi: 10.1016/s0387-7604(01)00263-7. PMID 11701251
- [Background] Luthvigsson P, Olafsson E, Sigurthardottir S, Hauser WA. Epidemiologic features of infantile spasms in Iceland. Epilepsia. 1994 Jul-Aug;35(4):802-5. doi: 10.1111/j.1528-1157.1994.tb02514.x. PMID 8082625
- [Background] Trevathan E, Murphy CC, Yeargin-Allsopp M. The descriptive epidemiology of infantile spasms among Atlanta children. Epilepsia. 1999 Jun;40(6):748-51. doi: 10.1111/j.1528-1157.1999.tb00773.x. PMID 10368073
- [Background] Hattori H. Spontaneous remission of spasms in West syndrome--implications of viral infection. Brain Dev. 2001 Nov;23(7):705-7. doi: 10.1016/s0387-7604(01)00278-9. PMID 11701282
- [Background] Hrachovy RA, Glaze DG, Frost JD Jr. A retrospective study of spontaneous remission and long-term outcome in patients with infantile spasms. Epilepsia. 1991 Mar-Apr;32(2):212-4. doi: 10.1111/j.1528-1157.1991.tb05246.x. PMID 1848513
- [Background] O'Callaghan FJ, Lux AL, Darke K, Edwards SW, Hancock E, Johnson AL, Kennedy CR, Newton RW, Verity CM, Osborne JP. The effect of lead time to treatment and of age of onset on developmental outcome at 4 years in infantile spasms: evidence from the United Kingdom Infantile Spasms Study. Epilepsia. 2011 Jul;52(7):1359-64. doi: 10.1111/j.1528-1167.2011.03127.x. Epub 2011 Jun 10. PMID 21668442
- [Background] Eisermann MM, DeLaRaillere A, Dellatolas G, Tozzi E, Nabbout R, Dulac O, Chiron C. Infantile spasms in Down syndrome--effects of delayed anticonvulsive treatment. Epilepsy Res. 2003 Jun-Jul;55(1-2):21-7. doi: 10.1016/s0920-1211(03)00088-3. PMID 12948613
- [Background] Jambaque I, Chiron C, Dumas C, Mumford J, Dulac O. Mental and behavioural outcome of infantile epilepsy treated by vigabatrin in tuberous sclerosis patients. Epilepsy Res. 2000 Feb;38(2-3):151-60. doi: 10.1016/s0920-1211(99)00082-0. PMID 10642043
- [Background] Pellock JM, Hrachovy R, Shinnar S, Baram TZ, Bettis D, Dlugos DJ, Gaillard WD, Gibson PA, Holmes GL, Nordl DR, O'Dell C, Shields WD, Trevathan E, Wheless JW. Infantile spasms: a U.S. consensus report. Epilepsia. 2010 Oct;51(10):2175-89. doi: 10.1111/j.1528-1167.2010.02657.x. PMID 20608959
- [Background] Mytinger JR, Joshi S; Pediatric Epilepsy Research Consortium, Section on Infantile Spasms. The current evaluation and treatment of infantile spasms among members of the Child Neurology Society. J Child Neurol. 2012 Oct;27(10):1289-94. doi: 10.1177/0883073812455692. Epub 2012 Aug 21. PMID 22914371
- [Background] Mackay MT, Weiss SK, Adams-Webber T, Ashwal S, Stephens D, Ballaban-Gill K, Baram TZ, Duchowny M, Hirtz D, Pellock JM, Shields WD, Shinnar S, Wyllie E, Snead OC 3rd; American Academy of Neurology; Child Neurology Society. Practice parameter: medical treatment of infantile spasms: report of the American Academy of Neurology and the Child Neurology Society. Neurology. 2004 May 25;62(10):1668-81. doi: 10.1212/01.wnl.0000127773.72699.c8. PMID 15159460
- [Background] Go CY, Mackay MT, Weiss SK, Stephens D, Adams-Webber T, Ashwal S, Snead OC 3rd; Child Neurology Society; American Academy of Neurology. Evidence-based guideline update: medical treatment of infantile spasms [RETIRED]. Report of the Guideline Development Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2012 Jun 12;78(24):1974-80. doi: 10.1212/WNL.0b013e318259e2cf. PMID 22689735
- [Background] Rho JM. Basic science behind the catastrophic epilepsies. Epilepsia. 2004;45 Suppl 5:5-11. doi: 10.1111/j.0013-9580.2004.05001.x. PMID 15283705
- [Background] Arya R, Shinnar S, Glauser TA. Corticosteroids for the treatment of infantile spasms: a systematic review. J Child Neurol. 2012 Oct;27(10):1284-8. doi: 10.1177/0883073812453203. Epub 2012 Aug 1. PMID 22859699
- [Background] Ben-Menachem E. Mechanism of action of vigabatrin: correcting misperceptions. Acta Neurol Scand Suppl. 2011;(192):5-15. doi: 10.1111/j.1600-0404.2011.01596.x. PMID 22061176
- [Background] Zhang B, McDaniel SS, Rensing NR, Wong M. Vigabatrin inhibits seizures and mTOR pathway activation in a mouse model of tuberous sclerosis complex. PLoS One. 2013;8(2):e57445. doi: 10.1371/journal.pone.0057445. Epub 2013 Feb 20. PMID 23437388
- [Background] Vanhatalo S, Nousiainen I, Eriksson K, Rantala H, Vainionpaa L, Mustonen K, Aarimaa T, Alen R, Aine MR, Byring R, Hirvasniemi A, Nuutila A, Walden T, Ritanen-Mohammed UM, Karttunen-Lewandowski P, Pohjola LM, Kaksonen S, Jurvelin P, Granstrom ML. Visual field constriction in 91 Finnish children treated with vigabatrin. Epilepsia. 2002 Jul;43(7):748-56. doi: 10.1046/j.1528-1157.2002.17801.x. PMID 12102679
- [Background] Westall CA, Nobile R, Morong S, Buncic JR, Logan WJ, Panton CM. Changes in the electroretinogram resulting from discontinuation of vigabatrin in children. Doc Ophthalmol. 2003 Nov;107(3):299-309. doi: 10.1023/b:doop.0000005339.23258.8f. PMID 14711162
- [Background] Simao GN, Zarei Mahmoodabadi S, Snead OC, Go C, Widjaja E. Abnormal axial diffusivity in the deep gray nuclei and dorsal brain stem in infantile spasm treated with vigabatrin. AJNR Am J Neuroradiol. 2011 Jan;32(1):199-203. doi: 10.3174/ajnr.A2224. Epub 2010 Aug 26. PMID 20801762
- [Background] Wheless JW, Carmant L, Bebin M, Conry JA, Chiron C, Elterman RD, Frost M, Paolicchi JM, Donald Shields W, Thiele EA, Zupanc ML, Collins SD. Magnetic resonance imaging abnormalities associated with vigabatrin in patients with epilepsy. Epilepsia. 2009 Feb;50(2):195-205. doi: 10.1111/j.1528-1167.2008.01896.x. Epub 2008 Nov 17. PMID 19054414
- [Background] Lux AL, Edwards SW, Hancock E, Johnson AL, Kennedy CR, Newton RW, O'Callaghan FJ, Verity CM, Osborne JP. The United Kingdom Infantile Spasms Study comparing vigabatrin with prednisolone or tetracosactide at 14 days: a multicentre, randomised controlled trial. Lancet. 2004 Nov 13-19;364(9447):1773-8. doi: 10.1016/S0140-6736(04)17400-X. PMID 15541450
- [Background] Jones K, Snead OC 3rd, Boyd J, Go C. Adrenocorticotropic hormone versus prednisolone in the treatment of infantile spasms post vigabatrin failure. J Child Neurol. 2015 Apr;30(5):595-600. doi: 10.1177/0883073814533148. Epub 2014 Jun 25. PMID 24965788
- [Background] Kossoff EH, Hartman AL, Rubenstein JE, Vining EP. High-dose oral prednisolone for infantile spasms: an effective and less expensive alternative to ACTH. Epilepsy Behav. 2009 Apr;14(4):674-6. doi: 10.1016/j.yebeh.2009.01.023. Epub 2009 Feb 4. PMID 19435579
- [Background] Ware TL, Mackay MT, Harvey AS, Freeman JL. Epileptic spasms: experience with a high-dose oral corticosteroid protocol. J Paediatr Child Health. 2012 Nov;48(11):985-9. doi: 10.1111/j.1440-1754.2012.02582.x. Epub 2012 Oct 8. PMID 23039949
- [Background] Hussain SA, Shinnar S, Kwong G, Lerner JT, Matsumoto JH, Wu JY, Shields WD, Sankar R. Treatment of infantile spasms with very high dose prednisolone before high dose adrenocorticotropic hormone. Epilepsia. 2014 Jan;55(1):103-7. doi: 10.1111/epi.12460. Epub 2013 Nov 8. PMID 24446954